CLINICAL TRIAL: NCT00790127
Title: A Multi-National, Blinded, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HQK-1001 in Subjects With Beta Thalassemia Intermedia, Including Hemoglobin E Beta Thalassemia
Brief Title: Phase 1/2 Study of HQK-1001 in Patients With Beta Thalassemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Susan Perrine, M.D. Chief Scientific Officer, VP Clinical Affairs, HemaQuest Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HQP-2008-003b
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- HQK-1001 (Experimental): HQK-1001
  Interventions: Drug: HQK-1001

INTERVENTIONS:
Drug: HQK-1001 — HQK-1001 capsules (10, 20, 30 or 40 mg) administered once a day, orally, for 56 days
  Arms: HQK-1001
Drug: Placebo — Matching placebo capsules administered once a day, orally, for 56 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of HQK-1001 administered daily for 8 weeks in subjects with beta thalassemia intermedia

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of beta thalassemia intermedia or hemoglobin E beta thalassemia
* Average of the initial two hemoglobin levels of less than 10 g/dL within ≥ 30 days prior to randomization.
* Age ≥ 12 and ≤ 60 years
* Able and willing to give informed consent or assent (if less than 18 years of age) and comply with all study procedures
* If female and of childbearing potential, must have a documented negative pregnancy test at Day -1 and must agree to use one or more locally medically accepted methods of contraception in the month prior to randomization, through the entire study, and for 4 weeks after the last dosing of study medication

Exclusion Criteria:

* Spleen palpable ≥ 2 cm below the left costal margin
* Pulmonary hypertension requiring oxygen therapy
* QTc > 450 msec on screening ECG
* Infection with hepatitis C, hepatitis B requiring therapy
* Known infection with HIV
* Red blood cell (RBC) transfusions within 2 months prior to administration of study medication with stable hemoglobin levels
* Fever greater than 38.5°C in the week prior to administration of study medication
* ALT > 4x upper limit of normal (ULN)
* Baseline elevation of CPK value prior to randomization
* Treatment with hydroxyurea within 2 months prior to administration of study medication
* Cancer diagnosis within 5 years of randomization (except for non-melanoma cutaneous malignancies)
* Serum creatinine > 1.5 mg/dl
* Received investigational systemic therapy within 30 days prior to randomization
* Currently pregnant or breast feeding a child
* Subject history of clinically significant arrhythmias or syncope
* Known current drug or alcohol abuse

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by (1) adverse events, (2) laboratory values (3) vital signs (4) physical exam | 168 days

SECONDARY OUTCOMES:
Pharmacokinetics assessed by plasma drug concentration levels | 140 days
Pharmacodynamics assessed by red blood cell production and induction of fetal hemoglobin | 168 days

CONTACTS AND LOCATIONS:
Overall Officials: Noppadol Siritanaratkul, MD, Principal Investigator — Siriraj Hospital
Locations (2):
- Chronic Care Center, Beirut, Lebanon
- Siriraj Hospital, Bangkok, Bangkoknoin District, Thailand

REFERENCES:
- [Derived] Foong WC, Loh CK, Ho JJ, Lau DS. Foetal haemoglobin inducers for reducing blood transfusion in non-transfusion-dependent beta-thalassaemias. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD013767. doi: 10.1002/14651858.CD013767.pub2. PMID 36637054